CLINICAL TRIAL: NCT04550624
Title: A Single Arm Phase II Study of Pembrolizumab in Combination With Lenvatinib in Patients With Advanced Biliary Tract Carcinoma After Progression on Standard Systemic Therapy
Brief Title: Pembrolizumab in Combination With Lenvatinib in Patients With Advanced Biliary Tract Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiahui International Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0001
Record Dates: First submitted 2020-08-31; First posted 2020-09-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Advanced Biliary Tract Carcinoma
Keywords: Advanced Biliary Tract Carcinoma; Pembrolizumab; Lenvatinib
MeSH Terms: interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional Arm (Experimental): This is an open-label, multi-center, phase II trial of lenvatinib in combination with pembrolizumab in patients with Advanced Biliary Tract Carcinoma (BTC) who have progressed on standard systemic therapy. All participants will be administered Pembrolizumab 200mg IV on day 1 and Lenvatinib 20mg PO daily days 1-21 of each cycle (21 days).
  Interventions: Drug: Pembrolizumab Injection [Keytruda]; Drug: Lenvatinib Mesylate

INTERVENTIONS:
Drug: Pembrolizumab Injection [Keytruda] — 200mg IV on day 1 of each cycle
  Other Names: Keytruda
Drug: Lenvatinib Mesylate — 20mg PO daily days 1-21 of each cycle
  Other Names: Lenvima

SUMMARY:
The prognosis for unresectable and metastatic biliary tract cancers (BTCs) including cholangiocarcinoma is poor with first line gemcitabine and cisplatin offering a median overall survival of 11.7 months. There is no standard second- or third-line therapy for advanced BTC, and this represents an unmet medical need for novel therapies. The immune system plays a critical role in the development of Advanced Biliary Tract Carcinoma (BTC) and chronic inflammation is a common underlying risk factor for BTC. Vascular endothelial growth factor (VEGF) signaling in BTC may lead to an immune suppression via inadequate tumor antigen presentation and an impaired T cell-mediated immune response directed against tumor antigens. Lenvatinib significantly decreased the population of immunosuppressive tumor-associated macrophages and increased interferon-γ-producing cluster of differentiation 8+ (CD8+) T cells. Addition of programmed cell death protein 1 (PD-1)/programmed death-ligand (PD-L1) inhibitors helps reverse VEGF-mediated immune suppression, restore T cell function, and promote T cell tumor infiltration. The combination of lenvatinib and pembrolizumab has demonstrated promising activity with manageable adverse events in various solid tumor types.

The investigators will assess the efficacy and safety of the combination of pembrolizumab and lenvatinib in patients with advanced BTC who failed standard therapy in this phase II study.

DETAILED DESCRIPTION:
Title: A Single Arm Phase II Study of Pembrolizumab in combination with Lenvatinib in Patients with Advanced Biliary Tract Carcinoma after Progression on Standard Systemic Therapy Study Description: The prognosis for unresectable and metastatic biliary tract cancers (BTCs) including cholangiocarcinoma is poor with first line gemcitabine and cisplatin offering a median overall survival of 11.7 months. There is no standard second- or third-line therapy for advanced BTC, and this represents an unmet medical need for novel therapies. The immune system plays a critical role in the development of Advanced Biliary Tract Carcinoma (BTC) and chronic inflammation is a common underlying risk factor for BTC. VEGF signaling in BTC may lead to an immune suppression via inadequate tumor antigen presentation and an impaired T cell-mediated immune response directed against tumor antigens. Lenvatinib significantly decreased the population of immunosuppressive tumor-associated macrophages and increased interferon-γ-producing CD8+ T cells. Addition of PD-1/PD-L1 inhibitors helps reverse VEGF-mediated immune suppression, restore T cell function, and promote T cell tumor infiltration. The combination of lenvatinib and pembrolizumab has demonstrated promising activity with manageable adverse events in various solid tumor types.

The investigators will assess the efficacy and safety of the combination of pembrolizumab and lenvatinib in patients with advanced BTC who failed standard therapy in this phase II study.

Objectives and Endpoints:

Primary Objective: Evaluate the objective response rate (ORR) (RECIST1.1) of lenvatinib in combination with pembrolizumab in patients with advanced BTC after progression on standard systemic therapies Secondary Objective: Evaluate the safety and tolerability of lenvatinib+pembrolizumab in this population; Determine the duration of response (DOR), progression free survival (PFS), and overall survival (OS); Determine the ORR, PFS and OS of subgroups stratified by molecular signatures (tumor mutation burden, PD-L1 expression, microsatellite instability (MSI) status, isocitrate dehydrogenase (IDH) or FGFR mutation/fusion status) in a pre-planned post-hoc analysis; Define molecular correlates of response, including circulating biomarkers and tumor tissue biomarkers Study Population: The study will enroll 40 patients who have unresectable or metastatic, histologically-confirmed advanced BTC. Both male and female patients age of 18 years or older who have failed standard systemic therapy for advanced BTC with measurable disease, adequate bone marrow reserve and hepatic/renal function, and ECOG performance status (PS) 0-1 could be eligible to participate in the study after completing the study enrollment screening tests and procedures.

Phase: II Description of Sites/Facilities Enrolling Participants: The study will be conducted at Jiahui International Cancer Center, Shanghai Jiahui International Hospital, in collaboration with Zhongshan Hospital.

Study treatment/Intervention: Each cycle is defined as 21 days treatment of Pembrolizumab in combination with Lenvatinib. Treatment will be administered on an outpatient basis:

Pembrolizumab 200mg IV day 1 of every 21 day-cycles; Lenvatinib 20mg PO once daily for 21-day cycles Study Duration: 24-36 months Participant Duration: up to 24 months

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the following criteria in order to be eligible to participate in the study:

  1. Unresectable or metastatic, histologically-confirmed advanced BTC (excluding periampullary cancer)
  2. Failed standard systemic therapy for advanced BTC due to progression of disease or toxicity
  3. Measurable disease
  4. Prior chemoembolization, radiofrequency ablation, or radiation to the liver is allowed as long as the patient has measurable disease outside the chemoembolization or radiation area or measurable progression at the site of chemoembolization or radiation
  5. ECOG Performance status ≤ 1
  6. Life expectancy > 3 months
  7. Adequate renal function as defined by Cr ≤ 1.5 upper limit of normal (ULN) or glomerular filtration rate (GFR) ≥ 60 mL/min/1.73 m2
  8. Adequate hepatic function as defined by bilirubin ≤ 2.5 x ULN and alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 5x ULN
  9. Adequate bone marrow reserve as evidenced by ANC > 1500/mcl, Plts >75,000/mcl, Hgb ≥ 9.0g/dl
  10. Prothrombin time / Partial thromboplastin time (PT/PTT) <1.5x ULN
  11. Urine Protein: Creatinine ratio of <1, if protein is > 2+ on urinalysis
  12. Age ≥ 18 years
  13. Participants with past or ongoing hepatitis C virus (HCV) infection are eligible for the study. Treated participants must have completed their treatment at least 1 month prior to starting study intervention. Untreated or incompletely treated HCV participants may initiate anti-viral therapy for HCV if liver function remains stable for at least 3 months on study intervention
  14. Participants with controlled hepatitis B are eligible for the study, as long as they meet the following criteria:

      Participants with chronic hepatitis B virus (HBV) infection, defined as HBsAg positive and/or detectable HBV DNA, must be given antiviral therapy for HBV for at least 4 weeks prior to the first dose of study intervention and HBV viral load must be less than 100 IU/ml. prior to the first dose of study treatment. Participants on active HBV therapy with viral loads under 100 IU/ml. should stay on the same therapy throughout study intervention. Antiviral therapy after completion of study intervention should follow local guidelines.
  15. Participants with clinically resolved HBV infection, defined as HBsAg negative and anti-hepatitis B core antigen (HBc) positive, and who have an undetectable HBV viral load at screening should be checked every 6 weeks for HBV viral load and treated for HBV if viral load is over 100 IU/ml. Antiviral therapy after completion of study intervention should follow local guidelines.

Exclusion Criteria:

* Patients who exhibit any of the following conditions at screening will not be eligible to be enrolled to the study:

  1. Prior treatment with other VEGF-R directed therapies
  2. Periampullary cancer
  3. Major surgery or radiation within the 4 weeks prior to enrollment; is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of registration. The treated patients must recover from their relevant treatment(i.e. to≤1 grade or baseline) and from any AEs caused by any previous treatment
  4. Uncontrolled hypertension defined by systolic blood pressure (SBP)>150 or diastolic blood pressure (DBP)>90 despite titration of anti-hypertensive medications
  5. Active, known or suspected autoimmune disease
  6. Congestive heart failure or symptomatic coronary artery disease within 3 months prior to enrollment
  7. Cerebrovascular accident within prior 6 months
  8. Clinically significant hemorrhage, bleeding event, or thromboembolic disease within six months
  9. History of bowel perforation
  10. History of (non-infectious) pneumonitis that required steroids or currently has pneumonitis
  11. Known history of HIV infection
  12. Severely impaired lung function or history of interstitial lung disease
  13. Concurrent malignancy (other than adequately treated non-melanoma skin cancer, superficial transitional cell carcinoma of the bladder, and cervical CIS) diagnosed within the past 5 years or any currently active malignancy
  14. Positive serum pregnancy test within 72 hours of first dosing of study treatment
  15. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of ORR | up to 36 months
  Evaluate the objective response rate (ORR) (RECIST1.1) of lenvatinib in combination with pembrolizumab in patients with advanced BTC after progression on standard systemic therapies

SECONDARY OUTCOMES:
All participants who receive at least one dose of study treatment will be evaluable for safety and tolerability through the monitoring of serious and non serious AEs, defined and graded according to NCI CTCAE v5.0. | up to 36 months
  All participants who receive at least one dose of study treatment will be evaluable for safety and tolerability in this study through the monitoring of all serious and non serious AEs, defined and graded according to NCI CTCAE v5.0 from the time of their first treatment.
Duration of Overall Response (DOR) | up to 36 months
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrence or PD is objectively documented, taking as reference for PD the smallest measurements recorded since the treatment started. Patients who do not relapse will be censored at the day of their last tumor assessment.
Progression-Free Survival (PFS) | up to 36 months
  Progression-Free Survival (PFS) is defined as the duration of time from start of treatment to time of objective disease progression or death from any cause without evidence of disease progression, whichever comes first.
Overall Survival (OS) | up to 36 months
  Overall Survival (OS) is defined as the duration of time from start of treatment to time of death.
Objective Response Rate (ORR) of subgroups burden | up to 36 months
  Determine the ORR of subgroups stratified by molecular signatures (tumor mutation burden, PD-L1 expression, MSI status, FGFR mutation/fusion status) in a pre-planned post-hoc analysis
Progression-Free Survival (PFS) of subgroups burden | up to 36 months
  Determine the PFS of subgroups stratified by molecular signatures (tumor mutation burden, PD-L1 expression, MSI status, FGFR mutation/fusion status) in a pre-planned post-hoc analysis
Overall Survival (OS) of subgroups burden | up to 36 months
  Determine the OS of subgroups stratified by molecular signatures (tumor mutation burden, PD-L1 expression, MSI status, FGFR mutation/fusion status) in a pre-planned post-hoc analysis

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Zhu, PhD, Principal Investigator — Shanghai JIH international Hospital
Locations (2):
- China (2):
  - Shanghai Jiahui International Hospital, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No